CLINICAL TRIAL: NCT07168161
Title: A Multicenter, Randomized, Double-Blind, Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of BDB-001 Injection in Patients With ANCA-Associated Vasculitis
Brief Title: BDB-001 Phase III Trial in ANCA-Associated Vasculitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STS-BDB001-10
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: ANCA Associated Vasculitis (AAV)
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — BDB001; Cyclophosphamide; Rituximab; Azathioprine; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BDB-001 injection group (Experimental): BDB-001 injection plus cyclophosphamide/azathioprine or rituximab plus prednisone-matching placebo.
  Interventions: Drug: BDB-001 injection; Drug: Cyclophosphamide; Biological: Rituximab; Drug: Azathioprine
- Prednisone group (Active Comparator): BDB-001 injection-matching placebo plus cyclophosphamide/azathioprine or rituximab plus a full starting dose of prednisone.
  Interventions: Drug: Cyclophosphamide; Biological: Rituximab; Drug: Azathioprine; Drug: Prednisone

INTERVENTIONS:
Drug: BDB-001 injection — Intravenously administered
  Arms: BDB-001 injection group
Drug: Cyclophosphamide — Intravenously administered
Biological: Rituximab — Intravenously administered
Drug: Azathioprine — Intravenously administered
Drug: Prednisone — Intravenously administered
  Arms: Prednisone group

SUMMARY:
The primary aim is to study the efficacy of treatment with BDB-001 Injection to induce remission in patients with active anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis (AAV), when used in combination with cyclophosphamide followed by azathioprine, or in combination with rituximab

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old≤Age≤75 years old, male or female;
2. Diagnosis of granulomatosis with polyangiitis(GPA) or microscopic polyangiitis(MPA)；
3. Newly diagnosed or relapsed GPA or MPA that requires treatment with a full starting dose of prednisone plus cyclophosphamide/azathioprine or rituximab；
4. Positive test for anti-proteinase 3(PR3) or anti-myeloperoxidase (MPO)；
5. Estimated glomerular filtration rate ≥15 mL/minute/1.73 m^2；
6. At least 1 major item, or at least 3 non-major items, or at least the 2 renal items on BVAS；

Exclusion Criteria:

1. Active tuberculosis infection;
2. alveolar hemorrhage requiring pulmonary ventilation support；
3. Any other known multi-system autoimmune disease including eosinophilic granulomatosis with polyangiitis (Churg-Strauss), systemic lupus erythematosus, IgA vasculitis (Henoch-Schönlein), rheumatoid vasculitis,anti-glomerular basement membrane disease, or cryoglobulinemic vasculitis；
4. HBsAg positive,or HBcAb positive and HBV-DNA positive；
5. Received CYC within 3 months before the first administration or Received rituximab(RTX) within 12 months before the first administration；
6. Received glucocorticoid shock therapy within 4 weeks before the first administration；
7. Received an oral daily dose of a GC of > 10 mg prednisone-equivalent for more than 6 weeks continuously before the first administration；
8. Received a anti-tumor necrosis factor and other biological agents treatment within 12 weeks before the first administration；
9. Received Continuous dialysis treatment for 12 weeks or more before the first administration; Received Dialysis within 1 week before the first administration;
10. Received intravenous immunoglobulin (Ig) or plasma exchange within 4 weeks before the first administration;
11. Pregnant or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2027-04-16 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieving disease remission assessed by Birmingham Vasculitis Activity Score (BVAS) | Week 24

SECONDARY OUTCOMES:
The proportion of patients achieving disease sustained remission assessed by Birmingham Vasculitis Activity Score (BVAS) | Week 48
Percentage of Subjects and Time to Experiencing a Relapse After Previously Achieving Remission in the Study | Week 48
Percentage of Participants With BVAS of 0 at Week 4 | Week 4
In Subjects With Renal Disease at Baseline (Based in the BVAS Renal Component), Change from baseline in Estimated glomerular filtration rate (eGFR) | Baseline, Week 24 and Week 48
In Subjects With Renal Disease at Baseline (Based in the BVAS Renal Component), Change from baseline in Urinary albumin:creatinine ratio (UACR) | Baseline, Week 4, 24 and 48
Glucocorticoid-induced Toxicity as Measured by Change From Baseline in the GTI | Baseline, Week 24 and 48
Cumulative dose of glucocorticoids | Week 24 and 48
Change from baseline in the Vasculitis Damage Index (VDI) | Baseline, Week 24 and 48
Change From Baseline in Health-related Quality of Life as Measured by the Domains and Component Scores of the SF-36 | Baseline, Week 24 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Minghui Zhao, M.D., Principal Investigator — Peking University First Hospital
Locations (50):
- China (50):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Shenzhen, Guangdong
  - Peking university Shenzhen Hospital, Shenzhen, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Guangxi Academy of Medical Sciences,The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi Zhuang Autonomous Region (gzar)
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The Second Hospital of Hebei Medical University City:Shijiazhuang, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Harbin, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital,Tongji Medical college of Hust, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - General Hospital of Hunan University of Medicine, Changde, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University (Nephrology Department), Changsha, Hunan
  - Xiangya Hospital Central South University(Rheumatism Immunity Branch), Changsha, Hunan
  - General Hospital of Hunan University of Medicine, Huaihua, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - Nanjing Gulou Hospital, Nanjing, Jiangsu
  - Nanjing University School of Medicine Affiliated Gulou Hospital, Nanjing, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Affiliated Hospital of Yanbian University (Yanbian Hospital), Yanbian, Jilin
  - Shengjing Hospital of China Medical University, Shengyang, Liaoning
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Neimenggu
  - Shandong Provincial Hospital, Jinan, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan hospital,Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xijing Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang